CLINICAL TRIAL: NCT05252429
Title: Phase ll Trial of Docetaxel/Pembrolizumab Combination Treatment in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Docetaxel/Pembrolizumab in Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hokkaido University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yasushi Shimizu, Clinical associate professor, Hokkaido University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020-011
Record Dates: First submitted 2022-02-03; First posted 2022-02-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: Effect of Drug
Keywords: head and neck cancer, docetaxel, pembrolizumab
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Docetaxel plus pembrolizumab (Experimental): Docetaxel 75mg/m2 plus pembrolizumab 200mg will be administered every 3 weeks intravenously for 6 cycles. Thereafter pembrolizumab 200mg every 3 weeks will be given as maintenance therapy until progression or up to 35 cycles.
  Interventions: Drug: Docetaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2; q21
  Other Names: Taxotere
Drug: Pembrolizumab — Pembrolizumab 200mg, q21
  Other Names: Keytruda

SUMMARY:
Pembrolizumab monotherapy and platinum-based chemotherapy in the combination with pembrolizumab for recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC) have been widely used in daily clinical practice based on the KEYNOTE-048 study. On the other hand, docetaxel is a commonly used antimitotic agent in cancer therapy and might have potent antitumor effect by the immune response. A combination therapy of docetaxel and pembrolizumab might be a promising treatment for R/M HNSCC. The KEYNOTE-048 study showed that pembrolizumab plus platinum and 5-fluorouracil is a tolerable treatment for R/M HNSCC. The main grade 3/4 adverse event of platinum and 5-fluorouracil was myelosuppression such as neutropenia similar to docetaxel in some studies for R/M HNSCC. The safety profile of platinum and 5-fluorouracil is not much different from docetaxel. Therefore, docetaxel/pembrolizumab combination treatment might also be tolerable. The hypothesis of this study is that a combination therapy of docetaxel and pembrolizumab will provide benefit for patients with R/M HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically-confirmed R/M HNSCC that is considered incurable by local therapies.

   Subjects should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was completed more than 6 months prior to signing consent if given as part of multimodal treatment for locally advanced disease is allowed.

   The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx. Subjects may not have a primary tumor site of nasopharynx (any histology).
2. Be willing and able to provide written informed consent for the trial.
3. Have results from testing of PD-L1 status.
4. Be ≥ 20 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have a performance status of 0 or 1 on the ECO G Performance Scale.
7. Have adequate organ function.
8. Have results from testing of HPV status for oropharyngeal cancer.
9. Female subjects of childbearing potential should have a negative blood pregnancy test within 72 hours prior to receiving the first dose of study medication.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy.

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent.
2. Has a life expectancy of less than 3 months and/ or has rapidly progressing disease in the opinion of the treating investigator.
3. Has received prior systemic anti-cancer therapy including radiation therapy, other non-systemic therapy or investigational agents within 4 weeks prior to the first dose of trial treatment.
4. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, or used an investigational device, any of which occurred within 4 weeks of the first dose of treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (using prednisolone ≥ 10mg per day) or any other form of immunosuppressive therapy within 7 days prior to the first dos e of trial treatment.
6. Has a diagnosed and/or treated additional malignancy within 2 years prior to randomization with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, curatively resected esophageal cancer, curatively resected in situ cervical cancer, and curatively resected in situ cancer.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
9. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis. Pneumonitis include active radiation pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has received prior therapy with an anti-PD-1, a nti-PD-L1, or anti-CTLA-4 agent.
12. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 year
  Overall response rate is estimated per RECIST 1.1 by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  For overall survival, the survival curve is estimated by the Kaplan-Meier method.
Progression-free survival (PFS) | 1 year
  For progression-free survival, the survival curve is estimated by the Kaplan-Meier method.
Duration of response (DoR) | 1 year
  For duration of response, the survival curve is estimated by the Kaplan-Meier method.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From treatment start date to 30 days after the final administration of the study drug
  Drug induced toxicities are assessed and graded according to Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yasushi Shimizu, Principal Investigator — Hokkaido University Hospital
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No